CLINICAL TRIAL: NCT00772525
Title: A Double-blind, Placebo-controlled, Randomized Crossover, Activity Study of Single Oral Doses of 50 mg and 400 mg Nerispirdine on Visual Function in Patients With Multiple Sclerosis
Brief Title: Single Oral Doses Study of Nerispirdine on Visual Function in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT10573
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Sclerosis; Optic Nerve; Neuritis
Keywords: Visual acuity; Contrast sensitivity; Visual Evoked Potentials; Optical Coherence Tomography
MeSH Terms: conditions — Multiple Sclerosis; Neuritis | interventions — nerispirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sequence 1 (Experimental): placebo,1 day treatment period 1
  50 mg Nerispirdine, 1 day treatment period 2
  400 mg Nerispirdine, 1 day treatment period 3
  Interventions: Drug: Nerispirdine; Drug: Placebo
- Sequence 2 (Experimental): placebo,1 day treatment period 1
  400 mg Nerispirdine, 1 day treatment period 2
  50 mg Nerispirdine, 1 day treatment period 3
  Interventions: Drug: Nerispirdine; Drug: Placebo
- Sequence 3 (Experimental): 50 mg Nerispirdine, 1 day treatment period 1
  placebo, 1 day treatment period 2
  400 mg Nerispirdine, 1 day treatment period 3
  Interventions: Drug: Nerispirdine; Drug: Placebo
- Sequence 4 (Experimental): 50 mg Nerispirdine, 1 day treatment period 1
  400 mg Nerispirdine, 1 day treatment period 2
  placebo, 1 day treatment period 3
  Interventions: Drug: Nerispirdine; Drug: Placebo
- Sequence 5 (Experimental): 400 mg Nerispirdine, 1 day treatment period 1
  placebo, 1 day treatment period 2
  50 mg Nerispirdine, 1 day treatment period 3
  Interventions: Drug: Nerispirdine; Drug: Placebo
- Sequence 6 (Experimental): 400 mg Nerispirdine, 1 day treatment period 1
  50 mg Nerispirdine, 1 day treatment period 2
  placebo, 1 day treatment period 3
  Interventions: Drug: Nerispirdine; Drug: Placebo

INTERVENTIONS:
Drug: Nerispirdine — form: tablet
  Route: oral
  Other Names: HP184
Drug: Placebo — form: tablet
  Route: oral

SUMMARY:
The primary objective of the study was to evaluate the effect of Nerispirdine (50 mg or 400 mg) and placebo given orally as a single dose once a week in crossover design on latency of Visual Evoked Potentials (VEP) P100 in optic nerves.

Secondary objectives included evaluation of the effect of Nerispirdine on VEP amplitude and other visual parameters including visual acuity and contrast, as well as evaluation of the safety and tolerability of Nerispirdine in patients with Multiple Sclerosis (MS).

Contrast sensitivity and visual acuity examinations (in addition to Optical Coherence Tomography [OCT] and VEPs) were needed during the screening period for defining etiologic relationships (if non-MS related impairment) and for assessing the effect of treatment of age-related eye disease versus the MS-related vision impairment.

DETAILED DESCRIPTION:
The crossover design included 3 treatment periods 1 week apart and 6 treatment sequences. Study participation were to be 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS (McDonald criteria), which includes patients with remitting-relapsing, secondary progressive, progressive-relapsing, or primary progressive MS who have had a past history of Optic Neuritis.

Exclusion Criteria:

* Multiple sclerosis exacerbation within 60 days of the Screening Visit and the relapse involved the visual fields or visual acuity
* No eye with appropriate degree of lesions for this study as defined by criteria based on degree of visual acuity deficit, refractive error, VEP P100 latency and average retinal nerve fiber layer thickness of as measured by Optical Coherence Tomography (OCT)
* Any MS-unrelated prior ophthalmological impairment (eg, compressive, ischemic, toxic, or nutritional optic neuropathies, Leber's hereditary optic atrophy)
* Previously exposed to 3,4-diaminopyridine or 4-aminopyridine

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Visual Evoked Potential (P100) latency | pre-dose and post-dose of each treatment intake (3)

SECONDARY OUTCOMES:
Pelli-Robson Contrast Sensitivity Score | pre-dose and post-dose of each treatment intake (3)
Early Treatment Diabetic Retinopathy Study (EDTRS) visual acuity score | pre-dose and post-dose of each treatment intake (3)
Visual Evoked Potential (VEP) amplitude | pre-dose and post-dose of each treatment intake (3)

CONTACTS AND LOCATIONS:
Overall Officials: Robert SERGOTT, MD, Principal Investigator — Wills Eye Institute, Thomas Jefferson University, Philadelphia Pennsylvania, USA
Locations (1):
- Sanofi-Aventis Administrave Office, Bridgewater, New Jersey, United States